CLINICAL TRIAL: NCT05422599
Title: A Randomised Double-blind Placebo-controlled Trial on Encapsulated Lemon Balm Efficacy and Tolerance on Sleep Quality Changes, and Mood and Wellbeing Effects Using Objective and Subjective Measures
Brief Title: Enhancement of Sleep Quality and Mood Following Supplementation With Lemon Balm in an Adult Population (Lemslp)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Naturex (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Chair of Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 22/01
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Sleep Disturbance; Mood Disturbance
Keywords: Sleep Quality, Sleep Onset Latency, Sleep Duration; Lemon Balm, Melissa Officinalis, Herbal Psychotropic; Sleep Diaries, Actiwatches, PSQI, Gut-Brain Axis Microbiota; Wellbeing, Antidepressant, Anxiolytic, Cognitive-Enhancing; Salivary Analytes, Melatonin, Cortisol
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — lemon balm leaf extract

STUDY DESIGN:
Intervention Model Description: Between and within groups model
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lemon balm (Experimental): 300mg Lemon balm and Maltodextrin
  Interventions: Dietary Supplement: Lemon balm
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lemon balm — 300mg Lemon balm and Maltoxdextrin capsules Other Name: Melissa Officinalis L.
  Arms: Lemon balm
Dietary Supplement: Placebo — 300mg Maltodextrin capsules
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of a 4-week dietary intervention of 300mg encapsulated aqueous lemon balm extract on measures of sleep quality, mood and well-being, alongside relevant biomarkers of circadian rhythms in healthy adults aged 18-40 years with mild sleep problems (PSQI entry of 5 and above). Three visits to the university alongside completing some home tests involving self-test stool, saliva and mood tests and wearing an wrist-secured actiwatch over 4-weeks whilst recording a daily sleep diary will be monitored to estimate sleep changes. Mood ratings, stool and saliva biomarkers will serve as a proxy to sleep improvement.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled, parallel-design study assessing the effect of a 4-week intervention of lemon balm extract (or matched placebo) in young to middle-age adults with mild sleep problems. A total of 108 participants will be randomly assigned to either 300 mg lemon balm extract or a matched placebo capsule consumed nightly before retiring to bed. The severity of sleep problems, depression, anxiety, perceived stress, quality of life and well-being will be measured at baseline and after 4 weeks of daily consumption. In addition, we will assess changes in microbiota and saliva neurohormone profiles at baseline and after 4 weeks of treatment.

Entry to the study to determine eligibility involves a sleep quality questionnaire (PSQI) score of 5 and above. The study comprises of a familiarisation visit and then two test days at the Nutritional Psychology Unit based at the University of Reading where primary sleep (PSQI), and exploratory measures of sleep (ISI, LSEQ) and mood (PANAS, Vivascentz(TM), FFS, PSS, DASS-21) tests will be completed. The screening visit will further assess habitual diet (Epic-Norfolk FFQ), and general health and lifestyle patterns to confirm eligibility. Participants will then continuously wear an wrist-secured actiwatch whilst recording a daily sleep diary to estimate sleep changes over the 4-week period. In addition, some further exploratory tests will be completed by participants from home 24h before baseline and 24h before post-intervention (saliva, stool, PANAS-X).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, between18-40 years old
* Mild Sleep problems (PSQI less than or equal to 5)
* Willingness to provide stool and saliva samples, wear an actiwatch and complete a nightly sleep diary.

Exclusion Criteria:

* Use medications that may affect the outcome
* Any long-term psychological or physiological health conditions
* Have any allergic reactions to ingredients in the capsules
* Have a BMI greater than or equal to 30
* Are vegetarian
* Taking any dietary supplements which they are unwilling to stop for the duration of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  A validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.

SECONDARY OUTCOMES:
Combined Sleep Diary and Research-Grade Actiwatch Sleep-Wake Patterns | Continuous over 4 weeks
  Passive motion tracking of sleep-wake patterns (heart rate variability) will be recorded via a wrist-worn research-grade actiwatch. The actiwatches will be secured on the participant's wrist throughout the study period. To cross-examine the actiwatch data, an in-house standardised daily sleep diary will measure sleep quality, sleep duration and sleep latency (how many times awoken during sleep time) (Carney et al., 2012; Orchard et al., 2020) where meaningful sleep outcomes will be manually inputted into actiwatch software at the end of sleep monitoring, as per standard practice in sleep research.
Diurnal Salivary Cortisol and Melatonin Patterns | 4 weeks
  Determination of changes in circadian sleep-wake patterns after 4-weeks daily 300mg lemon balm treatment by assessing diurnal sleep neurohormones, melatonin and cortisol. Changes in melatonin and cortisol will be assessed using 12 salivary self-test sampling kits taken in two windows (6 samples per window), within 24h before baseline day and within 24h before post-intervention day. For each test day, two samples will be taken first thing in the morning, 11am, 5pm and a final two samples in the evening. Sleep neurohormones will then be assessed against subjective sleep scores.
Gut Microbiota Changes | 4 weeks
  Examination of gut responses to mood and sleep physiology changes after 4-weeks daily 300mg lemon balm treatment by assessing changes in faecal microbiota levels. Two samples will be collected over the entire study. Microbiome diversity will be determined using self-test stool sampling kits taken in two windows, within 24h before baseline day and within 24h before post-intervention day. Faecal microbiota will then be compared to subjective sleep and mood scores.
Insomnia Severity Index (ISI) | 4 weeks
  A validated 7-item instrument designed to assess the nature, severity and impact of both nighttime and daytime components of insomnia within the last month. The scale ranges from 0 to 28 where higher scores indicate more severe insomnia.
Leeds Sleep Evaluation Questionnaire (LSEQ) | 4 weeks
  A 10-item self-report slider scale to evaluate ease of getting to sleep, sleep quality, ease of waking and behaviour following wakefulness. Higher scores indicate better sleep quality.
Perceived Stress Scale (PSS) | 4 weeks
  A validated 10-item questionnaire to measure levels of perceived stress. The scale ranges from 0 to 40 points with higher scores indicating greater stress levels.
Positive affect as measured by PANAS-X | 4 weeks
  General positive affect for assessing trait mood over the past month will be calculated by adding the values of 10 positive items in correspondence with the original PANAS, ranging from 0-50 where higher scores indicate positive affect. In addition, the expanded Positive and Negative Affect Schedule-X will assess higher order scales Surprise, Joviality,Self-Assurance, Attentiveness, and Serenity and these collective scores combined with general positive affect range from 0 to 170 points, where higher scores indicate better mood.
Positive affect as measured by PANAS-NOW | 4 weeks
  General positive affect for assessing transient mood as the respondent feels in the present moment will be calculated by adding the values of 10 positive items. Scores range from 0-50 points where higher scores indicate positive affect.
Negative affect as measured by PANAS-X | 4 weeks
  General positive affect for assessing trait mood over the past month will be calculated by adding the values of 10 negative items in correspondence with the original PANAS, ranging from 0-50 where higher scores indicate negative affect. In addition, the expanded Positive and Negative Affect Schedule-X will assess higher order scales Fear, Sadness, Guilt, Hostility, Shyness, Fatigue and these collective scores combined with general negative affect range from 0 to 170 points, where higher scores indicate worse mood.
Negative affect as measured by PANAS-NOW | 4 weeks
  General negative affect for assessing transient mood as the respondent feels in the present moment will be calculated by adding the values of 10 negative items, ranging from 0-50 where higher scores indicate negative affect.
Depression, Anxiety and Stress Scale - 21 items (DASS-21) | 4 weeks
  A validated 21-item measure to assess the severity of depression, anxiety and stress components, with 7 items per component. Each item is scored from 0-3 where higher scores indicate higher levels of distress in anxiety (scores range from 0 to >20), depression (0 to >28) and/or stress (0 to >34).
Flinders Fatigue Scale (FFS) | 4 weeks
  A self-report 7-item questionnaire to assess perception of frequency and severity of fatigue over the past 2 weeks. Global fatigue scores range from 0 to 31, where higher scores indicate greater fatigue.
Vivascentz(TM) Metric | 4 weeks
  An in-house Givaudan wellbeing metric, and patent approved (WO2020165463). This 18-item scale measures transient feelings in the present moment assessing 9 positive and 9 negative attributes (reverse scored) to contribute to overall wellbeing scores. Scores range from 0 to 180, where higher scores indicate higher wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, Professor, Principal Investigator — University of Reading
Locations (1):
- School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be made available on a platform such as Open Science Framework (www.osf.io) or a data repository linked to academic journals, in accordance with Open Science principles.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Scholey A, Gibbs A, Neale C, Perry N, Ossoukhova A, Bilog V, Kras M, Scholz C, Sass M, Buchwald-Werner S. Anti-stress effects of lemon balm-containing foods. Nutrients. 2014 Oct 30;6(11):4805-21. doi: 10.3390/nu6114805. PMID 25360512
- [Background] Araj-Khodaei M, Noorbala AA, Yarani R, Emadi F, Emaratkar E, Faghihzadeh S, Parsian Z, Alijaniha F, Kamalinejad M, Naseri M. A double-blind, randomized pilot study for comparison of Melissa officinalis L. and Lavandula angustifolia Mill. with Fluoxetine for the treatment of depression. BMC Complement Med Ther. 2020 Jul 3;20(1):207. doi: 10.1186/s12906-020-03003-5. PMID 32620104
- [Background] Kennedy DO, Scholey AB, Tildesley NT, Perry EK, Wesnes KA. Modulation of mood and cognitive performance following acute administration of Melissa officinalis (lemon balm). Pharmacol Biochem Behav. 2002 Jul;72(4):953-64. doi: 10.1016/s0091-3057(02)00777-3. PMID 12062586
- [Background] Haybar H, Javid AZ, Haghighizadeh MH, Valizadeh E, Mohaghegh SM, Mohammadzadeh A. The effects of Melissa officinalis supplementation on depression, anxiety, stress, and sleep disorder in patients with chronic stable angina. Clin Nutr ESPEN. 2018 Aug;26:47-52. doi: 10.1016/j.clnesp.2018.04.015. Epub 2018 May 19. PMID 29908682
- [Background] Ghazizadeh J, Hamedeyazdan S, Torbati M, Farajdokht F, Fakhari A, Mahmoudi J, Araj-Khodaei M, Sadigh-Eteghad S. Melissa officinalis L. hydro-alcoholic extract inhibits anxiety and depression through prevention of central oxidative stress and apoptosis. Exp Physiol. 2020 Apr;105(4):707-720. doi: 10.1113/EP088254. Epub 2020 Feb 21. PMID 32003913
- [Background] Noguchi-Shinohara M, Ono K, Hamaguchi T, Iwasa K, Nagai T, Kobayashi S, Nakamura H, Yamada M. Pharmacokinetics, Safety and Tolerability of Melissa officinalis Extract which Contained Rosmarinic Acid in Healthy Individuals: A Randomized Controlled Trial. PLoS One. 2015 May 15;10(5):e0126422. doi: 10.1371/journal.pone.0126422. eCollection 2015. PMID 25978046
- [Background] Buysse DJ, Hall ML, Strollo PJ, Kamarck TW, Owens J, Lee L, Reis SE, Matthews KA. Relationships between the Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), and clinical/polysomnographic measures in a community sample. J Clin Sleep Med. 2008 Dec 15;4(6):563-71. PMID 19110886
- [Background] Rivest RW, Schulz P, Lustenberger S, Sizonenko PC. Differences between circadian and ultradian organization of cortisol and melatonin rhythms during activity and rest. J Clin Endocrinol Metab. 1989 Apr;68(4):721-9. doi: 10.1210/jcem-68-4-721. PMID 2921307
- [Background] Carlson LE, Campbell TS, Garland SN, Grossman P. Associations among salivary cortisol, melatonin, catecholamines, sleep quality and stress in women with breast cancer and healthy controls. J Behav Med. 2007 Feb;30(1):45-58. doi: 10.1007/s10865-006-9082-3. Epub 2007 Jan 24. PMID 17245618
- [Background] Chang WP, Lin CC. Relationships of salivary cortisol and melatonin rhythms to sleep quality, emotion, and fatigue levels in patients with newly diagnosed lung cancer. Eur J Oncol Nurs. 2017 Aug;29:79-84. doi: 10.1016/j.ejon.2017.05.008. Epub 2017 Jun 2. PMID 28720269
- [Result] Ibarra A, Feuillere N, Roller M, Lesburgere E, Beracochea D. Effects of chronic administration of Melissa officinalis L. extract on anxiety-like reactivity and on circadian and exploratory activities in mice. Phytomedicine. 2010 May;17(6):397-403. doi: 10.1016/j.phymed.2010.01.012. Epub 2010 Feb 18. PMID 20171069
- [Result] Cases J, Ibarra A, Feuillere N, Roller M, Sukkar SG. Pilot trial of Melissa officinalis L. leaf extract in the treatment of volunteers suffering from mild-to-moderate anxiety disorders and sleep disturbances. Med J Nutrition Metab. 2011 Dec;4(3):211-218. doi: 10.1007/s12349-010-0045-4. Epub 2010 Dec 17. PMID 22207903
- [Result] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Result] Orchard F, Gregory AM, Gradisar M, Reynolds S. Self-reported sleep patterns and quality amongst adolescents: cross-sectional and prospective associations with anxiety and depression. J Child Psychol Psychiatry. 2020 Oct;61(10):1126-1137. doi: 10.1111/jcpp.13288. Epub 2020 Jun 17. PMID 32557672
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- See also: WHO (2002). World Health Organisation monographs on selected medicinal plants, Vol 2. — https://apps.who.int/iris/handle/10665/42052
- See also: Givaudan Vivascentz Wellbeing Metric — https://patentscope.wipo.int/search/en/detail.jsf?docId=WO2020165463&_cid=P22-KV9CB7-78639-1